CLINICAL TRIAL: NCT04612439
Title: Accuracy of Vacuum-assisted Breast Biopsy Elite 10G Versus BARD 14G Core Needle Biopsy of Abnormal Breast Lesions.
Brief Title: Accuracy of VABB Elite 10G Versus BARD 14G CNB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008222-12
Record Dates: First submitted 2020-09-14; First posted 2020-11-03 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VABB Elite 10G (Experimental): Vacuum-assisted Elite 10G
  Interventions: Device: VABB Elite 10G
- BARD 14G CNB (Active Comparator): BARD 14G Core needle
  Interventions: Device: BARD 14G CNB

INTERVENTIONS:
Device: VABB Elite 10G — If the biopsy device is a vacuum-assisted Elite 10G needle, insert the needle groove into the mass and rotate to cut the biopsy tissue one circle
  Arms: VABB Elite 10G
Device: BARD 14G CNB — If the biopsy device is a BARD 14G hollow core needle, insert the needle to the edge of the mass and pull the trigger in different directions to eject the needle to retrieve the material
  Arms: BARD 14G CNB

SUMMARY:
In this study, patients whose breast ultrasound showed a space-occupying lesion and needed biopsy to clarify the pathology were selected as the research subjects. This study aims to determine whether Vacuum-assisted biopsy device Elite is superior to the traditional BARD ejection type air core needle in the diagnosis of breast cancer through a prospective randomized study.

DETAILED DESCRIPTION:
The main purpose of the study was to analyze the difference in the accuracy of two biopsy devices in the diagnosis of breast cancer puncture. The purpose of the secondary study was to analyze the difference between the underestimation rate, false negative rate, sensitivity, and negative predictive value of the two devices, the consistency of the immunohistochemistry between the puncture pathology and surgical pathology of the two groups of patients, the number and time-consuming of the puncture acquisition specimens, and the two biopsies Differences in the incidence of complications (safety).

If the biopsy device is a vacuum-assisted Elite 10G needle, insert the needle groove into the mass and rotate to cut the biopsy tissue one circle; If the biopsy device is a BARD 14G hollow core needle, insert the needle to the edge of the mass and pull the trigger in different directions to eject the needle to retrieve the material.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old (including 18 years old)
* Ultrasound examination indicates the presence of space-occupying lesions in the breast. The size, location, and BI-RADS classification are not limited.
* Agree to undergo surgery after puncture
* Ability and willingness to sign informed consent

Exclusion Criteria:

* A biopsy has been performed in the external hospital
* Contraindications for puncture or surgery such as severe coagulation dysfunction
* Refuse breast surgery
* Axillary lymph node puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1470 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 3 months
  The accuracy of the puncture pathology was defined as the proportion of patients in the study population who were consistent with the qualitative diagnosis of the puncture pathology and surgical pathology.When the pathological diagnosis of puncture is "carcinoma in situ of the catheter", if the pathological diagnosis of the catheter is "carcinoma in situ of the catheter with microinfiltration", the puncture is considered accurate;If the surgical pathology confirms "invasive cancer (infiltrating lesion >1mm)", the pathology of the puncture is considered inaccurate (ie, underestimated)

SECONDARY OUTCOMES:
Concordance of immunohistochemical marker status | 3 months
  ER,PR, HER2and Ki67from tissues obtained by percutaneous biopsy and follow on surgical procedure.
Sensitivity | 3 months
  The proportion of patients with abreast cancer diagnosis by percutaneous biopsy among all patients receiving an invasive breast cancer diagnosis by either percutaneous biopsy or by follow on surgical procedure.
Negative Prediction Value | 3 months
  The proportion of patients whose diagnosis from percutaneous biopsy is benign, among all patients with a benign diagnosis by follow on surgical procedure, ORthe proportion of patients whose diagnosis from percutaneous biopsy is benign, among all patients whose malignant lesions were not diagnosed within less than 1 year of follow-up after initial percutaneous biopsy.
Underestimation Rate | 3 months
  The rate at which the surgical procedure following a percutaneous biopsy upgrades or upstages the severity of histopathologic diagnosis. For example, a) if percutaneous biopsy indicated benign lesions, and the subsequent surgical procedureidentifiedprecancerous lesions (e.g., ADH) or malignant lesions (DCIS or invasive adenocarcinoma); or b) if percutaneous biopsy indicated precancerous lesions, and follow up surgical procedureidentified malignant lesions(DCIS or invasive adenocarcinoma); or 3) if percutaneous biopsyindicated carcinoma in situ,and follow up surgical procedure identified infiltrating carcinoma (except microinvasive foci <1mm) identified by follow onsurgical procedure.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 7 days
  Rate of immediate bleeding on the day of puncture (bleeding requiring a compression bandage); rate of bleeding that cannot be stopped by a compression bandage within 48 hours after procedure; rate of hematoma on the second day after puncture; rate of skin ecchymosis and puncture point infection (local redness, swelling, heat and pain).

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Li, MD, Study Director — Fudan University; Ying Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Li J, Mo M, Shen J, Ren H, Li S, Liu G, Shao Z. The comparison of efficacy and safety evaluation of vacuum-assisted Elite 10-G system and the traditional BARD 14-G core needle in breast diagnosis: an open-label, parallel, randomized controlled trial. Int J Surg. 2023 May 1;109(5):1180-1187. doi: 10.1097/JS9.0000000000000257. PMID 37042316